CLINICAL TRIAL: NCT03675100
Title: Expression of Neurotrophic Factors, Tight Junction Proteins, and Cytokines According to the Irritable Bowel Syndrome Subtype and Sex
Brief Title: Neurotrophic Factors, Tight Junction Proteins, and Cytokines in IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B-1305/202-003
Record Dates: First submitted 2018-09-11; First posted 2018-09-18 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Irritable Bowel Syndrome; Tight Junction Alteration; Pathophysiology
Keywords: Irritable bowel syndrome; Subtype; Tight junction; Sex
MeSH Terms: conditions — Irritable Bowel Syndrome; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBS group (Sham Comparator): Patients who were diagnosed with IBS according to the ROME III criteria. Colonoscopic mucosal biopsy was undertaken for every subject.
  Interventions: Procedure: colonoscopic mucosal biopsy
- Control group (Active Comparator): Healthy participants who have no gastrointestinal symptoms and no colonoscopic abnormality. Colonoscopic mucosal biopsy was undertaken for every subject.
  Interventions: Procedure: colonoscopic mucosal biopsy

INTERVENTIONS:
Procedure: colonoscopic mucosal biopsy — colonoscopic mucosal biopsy was undertaken for every participant

SUMMARY:
To evaluate the role of neurotrophic factors (NGF, GDNF, TRPV-1), to quantity tight junction proteins (ZO-1, occludin, claudin) and cytokines (IL-8, TNF-a, IL-1b) in the colonic mucosa of IBS patients and also clarify sex differences in the pathophysiology of IBS.

ELIGIBILITY:
Inclusion Criteria:

* Control group Those who were between 18 and 80 years old and did not have any abnormalities in colonoscopy
* Irritable bowel syndrome group Patients who diagnosed as irritable bowel syndrome according to the ROME III criteria

Exclusion Criteria:

* history of IBD
* abdominal operation
* severe systemic disease
* malignancy,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
NGF, GDNF, and TRPV-1 mRNA expression of colonic mucosa | up to 24 weeks
  real-time qPCR

SECONDARY OUTCOMES:
ZO-1, Occludin, and Claudin mRNA expression of colonic mucosa | up to 24 weeks
  real-time qPCR and Western blot
IL-8, TNF-a, and IL-1b mRNA expression of colonic mucosa | up to 24 weeks
  real-time qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, Professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No